CLINICAL TRIAL: NCT04012112
Title: The Effect of Flexible Thoracolumbar Brace on Spinal Alignment, Pain and Quality of Life in Subjects With Neuromuscular Scoliosis : A Longitudinal Study
Brief Title: The Effect of Flexible Thoracolumbar Brace on Spinal Alignment, Pain and Quality of Life in Subjects With Neuromuscular Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-1807-481-005
Record Dates: First submitted 2019-06-05; First posted 2019-07-09 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Neuromuscular Scoliosis
Keywords: brace; neuromuscular disease; scoliosis
MeSH Terms: conditions — Neuromuscular Diseases; Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm trials (Experimental): longitudial study of the thoracolumbar brace in the neuromuscular scoliosis for 6 months
  Interventions: Device: thoracolumbar brace (Flexpine brace)

INTERVENTIONS:
Device: thoracolumbar brace (Flexpine brace) — Patient's would wear the FLEXpine brace over 18 hours a day for the 6 month

SUMMARY:
In the initial evaluation, the degree of spine is measured quantitatively using Cobb's angle and Muscular Dystrophy Spine Questionnaire (MDSQ). The patients who had Cobbs angle of 20-45 'by spinal plain radiography were evaluated for the effects of flexpine brace wearing and rehabilitation for 6 months. After 12 months, whole spine X-ray was taken for the followed up the patient's status.

ELIGIBILITY:
Inclusion Criteria:

* 20-45' degrees of cobb's angle in the neuromuscular disease

Exclusion Criteria:

* patient's who had spinal surgery
* less than 20 degree or more than 45 degree of cobb's angle
* acute lumbar pain

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
change of the scoliosis | 6months
  Cobb's angle in the whole spine anteroposterior view of X-ray before, immediately after, and 6-month after wearing FLEXpine brace

SECONDARY OUTCOMES:
change of pain | 6months
  pain scale checked through the visual analog scale
change of pulmonary function | 6 months
  assessed by spirometer of forced vical capacity
change of quality of life | 6 months
  Parents assessed the quality of life through the muscular dystrophy spine qusetionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Bundang, South Korea

IPD SHARING:
Plan to Share IPD: Undecided